CLINICAL TRIAL: NCT01757665
Title: ProspeCtive, nOn-randoMized, MulticENter Clinical Evaluation of Edwards Pericardial Aortic and Mitral Bioprostheses (Models 11000A and 11000M) With a New Tissue Treatment Platform (COMMENCE)
Brief Title: ProspeCtive, nOn-randoMized, MulticENter Clinical Evaluation of Edwards Pericardial Bioprostheses With a New Tissue Treatment Platform (COMMENCE)
Acronym: COMMENCE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-02
Record Dates: First submitted 2012-12-18; First posted 2012-12-31 (Estimated); Results first posted 2019-12-27 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Aortic Stenosis; Mitral Stenosis; Aortic Valve Insufficiency; Mitral Valve Insufficiency; Heart Failure
Keywords: Aortic valve replacement; Mitral valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis; Mitral Valve Stenosis; Aortic Valve Insufficiency; Mitral Valve Insufficiency; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Bioprosthesis: Aortic Model 11000A/ Mitral Model 11000M (Experimental): Aortic/Mitral valve replacement therapy
  Interventions: Device: Edwards Aortic and Mitral Bioprostheses Models 11000A and 11000M

INTERVENTIONS:
Device: Edwards Aortic and Mitral Bioprostheses Models 11000A and 11000M — Implant of an aortic valve, Model 11000A or mitral valve, Model 11000M

SUMMARY:
The objective of this trial is to confirm that the modifications to tissue processing, valve sterilization and packaging do not raise any new questions of safety and effectiveness in subjects who require replacement of their native or prosthetic aortic or mitral valve.

DETAILED DESCRIPTION:
Multicenter, prospective, single arm trial - Up to seven hundred (700) aortic valve replacement (AVR) subjects and up to one hundred seventy-five (175) mitral valve replacement (MVR) subjects at up to forty (40) clinical sites will be enrolled. The trial will include male and female patients, 18 years or older, requiring replacement for a diseased, damaged, or malfunctioning native or prosthetic aortic or mitral valve. Patients will be followed and assessed after implant for up to 5 years.

ELIGIBILITY:
Eligibility Criteria:

Inclusion Criteria:

1. Is 18 years or older
2. Provides written informed consent prior to trial procedures
3. Agrees to attend all follow-up assessments for up to 5 years and is willing to comply with specified follow-up evaluations at clinical investigational sites that are participating in the COMMENCE trial and/or obtain the protocol-specified diagnostic tests at centers that are under the same IRB or the same healthcare system
4. Diagnosed with aortic or mitral valve disease requiring valve replacement based on pre- operative evaluation
5. Scheduled to undergo planned aortic or mitral valve replacement with or without concomitant bypass surgery
6. Scheduled to undergo planned aortic valve replacement with or without resection and replacement of the ascending aorta from the sinotubular junction and without the need for circulatory arrest for hemi arch or arch replacement

Exclusion criteria:

A subject meeting any of the following criteria shall be excluded:

1. Requires emergency surgery
2. Requires planned multiple valve replacement/ repair (with the exception of mitral valve replacement with tricuspid valve repair)
3. Has prior valve surgery, which included implant of a bioprosthetic valve, mechanical valve, or annuloplasty ring that will remain in situ
4. Requires a surgical procedure outside of the cardiac area (e.g. vascular bypass)
5. Requires surgical replacement of the aortic root
6. Has active endocarditis/myocarditis or endocarditis/myocarditis within 3 months to the scheduled aortic or mitral valve replacement surgery
7. Has renal insufficiency as determined by creatinine (S-Cr) level ≥ 2.5 mg/dL or end -stage renal disease requiring chronic dialysis at screening visit
8. Has MRI or CT scan confirmed stroke, cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months (180 days) prior to planned valve surgery
9. Has acute myocardial infarction (MI) within 30 days prior to planned valve surgery
10. Has presence of non-cardiac disease limiting life expectancy to less than 12 months
11. Diagnosed with hypertrophic obstructive cardiomyopathy (HOCM)
12. Diagnosed with abnormal calcium metabolism and hyperparathyroidism
13. Exhibits left ventricular ejection fraction ≤ 20% as validated by diagnostic procedure prior to planned valve surgery
14. Echocardiographic evidence of an intra-cardiac mass, thrombus, or vegetation
15. Hemodynamic or respiratory instability requiring inotropic support, mechanical circulatory support, or mechanical ventilation within 30 days prior to planned valve surgery
16. Documented leukopenia (WBC < 3.5x 10³/μL), acute anemia (Hgb < 10.0 gm/dL or 6 mmol/L) or thrombocytopenia (platelet count < 50x 10³/μL) accompanied by history of bleeding diathesis and coagulopathy
17. Has prior organ transplant or is currently an organ transplant candidate
18. Current or recent participation (within 6 weeks prior to surgery) in another drug or device trial
19. Was previously implanted with trial device (Model 11000A or Model 11000M)
20. Pregnant (female subject of childbearing potential only), lactating or planning to become pregnant during the duration of participation in trial
21. Currently incarcerated or unable to give voluntary informed consent
22. Documented history of substance (drug or alcohol) abuse within the last 5 years prior to implant
23. Requires concomitant left ventricular assist device (LVAD) placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 777 (Actual)
Dates: Start 2012-12-11 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2026-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John Puskas, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (32):
- United States (29):
  - Cardiology, P.C., Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - Sutter Institute for Medical Research, Sacramento, California
  - Board of Trustees of the Leland Stanford Junior University, Stanford, California
  - Yale-New Haven, New Haven, Connecticut
  - Shands at the University of Florida, Gainesville, Florida
  - Florida Hospital, Orlando, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Spectrum Health Hospital, Grand Rapids, Michigan
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Washington University/ Barnes Jewish Hospital, St Louis, Missouri
  - New York Weill Cornell Medical Center, New York, New York
  - Mount Sinai Morningside, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - New York Presbyterian Hospital - Columbia University Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Pinnacle Health Cardiovascular Institute, Mechanicsburg, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - St. Thomas Health, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - The Heart Hospital of Baylor Plano, Plano, Texas
  - University of Utah, Salt Lake City, Utah
- Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Canada
- Poland (2):
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow
  - The Cardinal Stefan Wyszynski Institute of Cardiology, Warsaw

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.

REFERENCES:
- [Result] Puskas JD, Bavaria JE, Svensson LG, Blackstone EH, Griffith B, Gammie JS, Heimansohn DA, Sadowski J, Bartus K, Johnston DR, Rozanski J, Rosengart T, Girardi LN, Klodell CT, Mumtaz MA, Takayama H, Halkos M, Starnes V, Boateng P, Timek TA, Ryan W, Omer S, Smith CR; COMMENCE Trial Investigators. The COMMENCE trial: 2-year outcomes with an aortic bioprosthesis with RESILIA tissue. Eur J Cardiothorac Surg. 2017 Sep 1;52(3):432-439. doi: 10.1093/ejcts/ezx158. PMID 28605428
- [Result] Johnston DR, Griffith BP, Puskas JD, Bavaria JE, Svensson LG; COMMENCE Trial Investigators. Intermediate-term outcomes of aortic valve replacement using a bioprosthesis with a novel tissue. J Thorac Cardiovasc Surg. 2021 Nov;162(5):1478-1485. doi: 10.1016/j.jtcvs.2020.01.095. Epub 2020 Feb 21. PMID 32340804
- [Result] Bavaria JE, Griffith B, Heimansohn DA, Rozanski J, Johnston DR, Bartus K, Girardi LN, Beaver T, Takayama H, Mumtaz MA, Rosengart TK, Starnes V, Timek TA, Boateng P, Ryan W, Cornwell LD, Blackstone EH, Borger MA, Pibarot P, Thourani VH, Svensson LG, Puskas JD; COMMENCE Trial Investigators. Five-year Outcomes of the COMMENCE Trial Investigating Aortic Valve Replacement With RESILIA Tissue. Ann Thorac Surg. 2023 Jun;115(6):1429-1436. doi: 10.1016/j.athoracsur.2021.12.058. Epub 2022 Jan 20. PMID 35065065
- [Result] Heimansohn DA, Baker C, Rodriguez E, Takayama H, Dagenais F, Talton DS, Mumtaz MA, Pibarot P, Puskas JD; COMMENCE Trial Investigators. Mid-term outcomes of the COMMENCE trial investigating mitral valve replacement using a bioprosthesis with a novel tissue. JTCVS Open. 2023 Jun 2;15:151-163. doi: 10.1016/j.xjon.2023.05.008. eCollection 2023 Sep. PMID 37808026
- [Result] Beaver T, Bavaria JE, Griffith B, Svensson LG, Pibarot P, Borger MA, Sharaf OM, Heimansohn DA, Thourani VH, Blackstone EH, Puskas JD; COMMENCE Trial Investigators. Seven-year outcomes following aortic valve replacement with a novel tissue bioprosthesis. J Thorac Cardiovasc Surg. 2024 Sep;168(3):781-791. doi: 10.1016/j.jtcvs.2023.09.047. Epub 2023 Sep 29. PMID 37778503
- [Result] Bavaria JE, Mumtaz MA, Griffith B, Svensson LG, Pibarot P, Borger MA, Thourani VH, Blackstone EH, Puskas JD. Five-Year Outcomes After Bicuspid Aortic Valve Replacement With a Novel Tissue Bioprosthesis. Ann Thorac Surg. 2024 Jul;118(1):173-179. doi: 10.1016/j.athoracsur.2023.11.036. Epub 2023 Dec 21. PMID 38135262
- [Result] Thourani VH, Puskas JD, Griffith B, Svensson LG, Pibarot P, Borger MA, Heimansohn D, Beaver T, Blackstone EH, Antonio ALM, Bavaria JE; COMMENCE Trial Investigators. Five-year comparison of clinical and echocardiographic outcomes of pure aortic stenosis with pure aortic regurgitation or mixed aortic valve disease in the COMMENCE trial. JTCVS Open. 2024 Sep 10;22:160-173. doi: 10.1016/j.xjon.2024.08.020. eCollection 2024 Dec. PMID 39780838
- [Result] Salna M, Bavaria JE, Heimansohn D, Beaver T, Griffith B, Svensson LG, Pibarot P, Borger MA, Thourani VH, Blackstone EH, Cornwell LD, Puskas JD, Takayama H. Seven-Year Results for RESILIA Tissue in Bicuspid Aortic Valve Replacement Patients: Age and Valve Size Considerations. Interdiscip Cardiovasc Thorac Surg. 2025 Aug 5;40(8):ivaf176. doi: 10.1093/icvts/ivaf176. PMID 40748697
- See also: New York Heart Association Classification — https://www.heart.org/en/health-topics/heart-failure/what-is-heart-failure/classes-of-heart-failure
- See also: Short Form Health Survey (SF-12) — https://www.physio-pedia.com/12-Item_Short_Form_Survey_(SF-12)

RESULTS

PARTICIPANT FLOW:
Groups:
- Edwards Pericardial Aortic Bioprosthesis, Model 11000A: The Edwards Pericardial Aortic Bioprosthesis, Model 11000A, is indicated for patients who require replacement of their native or prosthetic aortic valve.
- Edwards Pericardial Mitral Bioprosthesis, Model 11000M: The Edwards Pericardial Mitral Bioprosthesis, Model 11000M, is indicated for patients who require replacement of their native or prosthetic mitral valve.
Period: Overall Study
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A | Edwards Pericardial Mitral Bioprosthesis, Model 11000M
Started | 694 | 83
Implanted With Device | 689 | 82
Completed | 0 | 0
Not Completed | 694 | 83
Not completed — Still on Study - Visit Completed | 240 | 30
Not completed — Still on Study - Visit Pending | 398 | 40
Not completed — Still on Study - Missed Visit | 14 | 1
Not completed — Death | 25 | 8
Not completed — Explant | 1 | 2
Not completed — Withdrawal by Subject | 10 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Not Implanted with Device | 5 | 1

BASELINE CHARACTERISTICS:
Population: This outcome is reported for enrolled subjects where data is available. Subjects were considered enrolled after meeting all the enrollment criteria, signing the informed consent, and after the surgeon assesses the subject's anatomy, sizes the annulus, and determines that the trial valve can be implanted.
Groups:
- Total: Total of all reporting groups
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A | Edwards Pericardial Mitral Bioprosthesis, Model 11000M | Total
Number analyzed (Participants) | 694 | 83 | 777
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (11.6) | 68.9 (9.3) | 67.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 49 | 245
  Male | 498 | 34 | 532
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 23 | 2 | 25
  White | 622 | 73 | 695
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 37 | 6 | 43

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Structural Valve Deterioration
Description: The rate of implanted subjects that experience structural valve deterioration (SVD) of the trial valve by the time of the post operative day (POD) 390 follow-up visit. Structural valve deterioration includes dysfunction or deterioration intrinsic to the valve. Examples of SVD includes complications such as wear, fracture, calcification, leaflet tear.
Time Frame: 1 Year Post Implant
Population: The outcome is reported for subjects who received the Model 11000A or Model 11000M device where data is available. The SVD result combines the aortic and mitral implanted subjects. The study was powered for the combined cohort for this endpoint as there would be too few mitral subjects to report the arms separately.
Measure: Count of Participants; unit: Participants
Groups:
- Edwards Pericardial Bioprosthesis, Models 11000A & 11000M: The Edwards Pericardial Aortic Bioprosthesis, Model 11000A, is indicated for patients who require replacement of their native or prosthetic aortic valve.
  The Edwards Pericardial Mitral Bioprosthesis, Model 11000M, is indicated for patients who require replacement of their native or prosthetic mitral valve.
Arm/Group | Edwards Pericardial Bioprosthesis, Models 11000A & 11000M
Number analyzed (Participants) | 716
Participants | 1
Statistical Analysis 1: Comparison: Edwards Pericardial Bioprosthesis, Models 11000A & 11000M; The null hypothesis is that the rate of structural valve deterioration at one year is greater than 1%. The alternative hypothesis is that this rate is less than 1%; Test type: Superiority; percent of patients = 0.1, 95% CI 1-sided [upper limit 0.7] — Upper 95% CI was calculated by the method of Clopper and Pearson, using the Beta distribution with parameters x + 1 and n - x where x is the number of SVD events by POD 390 and n is the number of subjects followed at the 1 year assessment

2. Secondary Outcome: Percentage of Subjects With Early Adverse Events
Description: Number of subjects with early adverse events occurring within 30 days of procedure divided by the number of enrolled subjects times 100
Time Frame: Events occuring within 30 days of procedure
Population: The outcome is reported for subjects who received the Model 11000A or Model 11000M device where data is available.
Measure: Number; unit: percentage of subjects
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A | Edwards Pericardial Mitral Bioprosthesis, Model 11000M
Number analyzed (Participants) | 689 | 82
percentage of subjects
  All Cause Mortality | 1.2 | 1.2
  Trial Valve Related Mortality | 0.4 | 1.2
  Thromboembolism | 2.2 | 2.4
  Valve Thrombosis | 0.0 | 0.0
  All Bleeding | 0.9 | 1.2
  Major Bleeding | 0.7 | 1.2
  Endocarditis | 0.0 | 0.0
  Hemolysis | 0.0 | 0.0
  All Paravalvular Leak (OPC) | 0.3 | 0.0
  Major Paravalvular Leak (OPC) | 0.1 | 0.0
  Non-structural Valve Dysfunction | 0.0 | 0.0
  Reoperation | 0.1 | 0.0
  Explant | 0.0 | 0.0

3. Secondary Outcome: Percentage of Late Adverse Events Divided by Late Patient Years
Description: Number of late events divided by the total number of late patient years times 100. Late patient years are calculated from 31 days post-implant to the date of the last contact (follow up or adverse event).
Time Frame: Events occurring >= 31 days and up through 3 years post-implant
Population: The outcome is reported for subjects who received the Model 11000A or Model 11000M device where data is available.
Measure: Number; unit: percentage of events/late patient years
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A | Edwards Pericardial Mitral Bioprosthesis, Model 11000M
Number analyzed (Participants) | 689 | 82
percentage of events/late patient years
  All Cause Mortality | 2.2 | 6.1
  Trial Valve Related Mortality | 0.7 | 0.9
  Thromboembolism | 2.1 | 1.7
  Valve Thrombosis | 0.0 | 0.0
  All Bleeding | 2.6 | 8.7
  Major Bleeding | 1.4 | 5.2
  Endocarditis | 0.6 | 0.9
  Hemolysis | 0.0 | 0.0
  All Paravalvular Leak (OPC) | 0.2 | 0.0
  Major Paravalvular Leak (OPC) | 0.1 | 0.0
  Non-structural Valve Dysfunction | 0.0 | 0.9
  Reoperation | 0.2 | 2.6
  Explant | 0.2 | 1.7

4. Other Pre Specified Outcome: Subject's Average Mean Gradient Measurements - 11000A
Description: Mean gradient is the average flow of blood through the aortic valve measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. Mean gradient values depend on the size and type of valve.
Time Frame: 3 Months, 1 Year, and 2 Year Post Implant
Population: The outcome is reported for subjects who received the Model 11000A device where data is available.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 19mm; Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 21mm; Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 23mm; Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 25mm; Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 27mm; Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 29mm; Edwards Pericardial Aortic Bioprosthesis, Model 11000A - Total: The Edwards Pericardial Aortic Bioprosthesis, Model 11000A, is indicated for patients who require replacement of their native or prosthetic aortic valve.
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 19mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 21mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 23mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 25mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 27mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 29mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - Total
Number analyzed (Participants) | 22 | 131 | 214 | 202 | 100 | 20 | 689
mmHg
  3 Months: number analyzed (Participants) | 22 | 118 | 196 | 185 | 90 | 12 | 623
  3 Months | 13.8 (6.1) | 10.7 (4.2) | 9.4 (3.8) | 8.7 (3.4) | 6.8 (2.6) | 4.7 (1.3) | 9.1 (4.0)
  1 Year: number analyzed (Participants) | 16 | 97 | 158 | 132 | 69 | 0 | 472
  1 Year | 17.6 (7.8) | 12.6 (4.7) | 10.1 (3.8) | 9.6 (5.2) | 8.2 (3.5) |  | 10.4 (4.9)
  2 Year: number analyzed (Participants) | 8 | 42 | 66 | 49 | 17 | 0 | 182
  2 Year | 16.1 (6.4) | 11.2 (4.0) | 9.9 (4.4) | 9.2 (3.4) | 8.3 (3.5) |  | 10.1 (4.3)

5. Other Pre Specified Outcome: Subject's Average Mean Gradient Measurements - 11000M
Description: Mean gradient is the average flow of blood through the mitral valve measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. Mean gradient values depend on the size and type of valve.
Time Frame: 3 Months, 1 Year, and 2 Years Post Implant
Population: The outcome is reported for subjects who received the Model 11000M device where data is available.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 25mm; Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 27mm; Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 29mm; Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 31mm; Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 33mm; Edwards Pericardial Mitral Bioprosthesis, Model 11000M - Total: The Edwards Pericardial Mitral Bioprosthesis, Model 11000M, is indicated for patients who require replacement of their native or prosthetic mitral valve.
Arm/Group | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 25mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 27mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 29mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 31mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 33mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - Total
Number analyzed (Participants) | 6 | 29 | 25 | 16 | 6 | 82
mmHg
  3 Months: number analyzed (Participants) | 5 | 26 | 23 | 14 | 6 | 74
  3 Months | 5.6 (0.7) | 4.1 (1.7) | 4.0 (1.5) | 3.4 (1.3) | 3.3 (1.4) | 4.0 (1.6)
  1 Year: number analyzed (Participants) | 4 | 25 | 20 | 12 | 6 | 67
  1 Year | 4.9 (1.2) | 4.1 (1.4) | 4.1 (1.5) | 3.9 (2.0) | 3.3 (1.4) | 4.0 (1.5)
  2 Year: number analyzed (Participants) | 0 | 13 | 6 | 2 | 2 | 23
  2 Year |  | 3.9 (1.8) | 3.8 (1.0) | 3.5 (0.8) | 3.4 (2.5) | 3.8 (1.5)

6. Other Pre Specified Outcome: Subject's Average Peak Gradients Measurements Over Time - 11000A
Description: Peak gradient is the maximum value measured of flow of blood through the aortic valve as measured in millimeters of mercury. Gradients are evaluated by echocardiography over time.
Time Frame: 3 Months, 1 Year, and 2 Years Post Implant
Population: The outcome is reported for subjects who received the Model 11000A device where data is available.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 19mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 21mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 23mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 25mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 27mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 29mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - Total
Number analyzed (Participants) | 22 | 131 | 214 | 202 | 100 | 20 | 689
mmHg
  3 Month: number analyzed (Participants) | 22 | 118 | 196 | 185 | 90 | 12 | 623
  3 Month | 27.5 (12.3) | 21.7 (8.2) | 18.8 (6.9) | 17.5 (6.3) | 13.8 (4.9) | 10.1 (3.0) | 18.4 (7.6)
  1 Year: number analyzed (Participants) | 16 | 97 | 158 | 132 | 69 | 0 | 472
  1 Year | 35.0 (16.3) | 25.2 (8.9) | 20.1 (7.5) | 19.2 (8.9) | 16.7 (6.9) |  | 20.9 (9.3)
  2 Year: number analyzed (Participants) | 8 | 42 | 66 | 49 | 17 | 0 | 182
  2 Year | 31.7 (12.0) | 22.0 (7.5) | 19.8 (8.5) | 18.2 (6.0) | 16.4 (6.6) |  | 20.1 (8.2)

7. Other Pre Specified Outcome: Subject's Average Peak Gradients Measurements Over Time - 11000M
Description: Peak gradient is the maximum value measured of flow of blood through the mitral valve as measured in millimeters of mercury. Gradients are evaluated by echocardiography over time.
Time Frame: 3 Months, 1 Year, and 2 Years Post Implant
Population: The outcome is reported for subjects who received the Model 11000M device where data is available.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 25mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 27mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 29mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 31mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 33mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - Total
Number analyzed (Participants) | 6 | 29 | 25 | 16 | 6 | 82
mmHg
  3 Months: number analyzed (Participants) | 5 | 26 | 23 | 14 | 6 | 74
  3 Months | 12.0 (1.4) | 9.8 (4.0) | 10.2 (4.2) | 9.0 (2.8) | 17.4 (22.1) | 10.5 (7.1)
  1 Year: number analyzed (Participants) | 4 | 25 | 20 | 12 | 6 | 67
  1 Year | 10.6 (3.0) | 9.9 (3.2) | 10.4 (3.7) | 10.2 (5.5) | 9.0 (4.1) | 10.1 (3.8)
  2 Year: number analyzed (Participants) | 0 | 13 | 6 | 2 | 2 | 23
  2 Year |  | 9.5 (4.7) | 10.5 (3.4) | 6.6 (1.2) | 8.3 (3.4) | 9.4 (4.0)

8. Other Pre Specified Outcome: Subject's Average Effective Orifice Area Measurements - 11000A
Description: Effective orifice area represents the cross-sectional area of the blood flow downstream of the aortic valve. Effective orifice area is evaluated by echocardiography over time.
Time Frame: 3 Months, 1 Year, and 2 Years Post Implant
Population: The outcome is reported for subjects who received the Model 11000A device where data is available.
Measure: Mean (Standard Deviation); unit: Centimeters Squared
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 19mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 21mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 23mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 25mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 27mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 29mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - Total
Number analyzed (Participants) | 22 | 131 | 214 | 202 | 100 | 20 | 689
Centimeters Squared
  3 Months: number analyzed (Participants) | 22 | 117 | 196 | 184 | 90 | 11 | 620
  3 Months | 1.4 (0.4) | 1.5 (0.4) | 1.7 (0.4) | 1.8 (0.5) | 2.3 (0.7) | 2.5 (0.8) | 1.8 (0.6)
  1 Year: number analyzed (Participants) | 16 | 97 | 155 | 131 | 68 | 0 | 467
  1 Year | 1.1 (0.2) | 1.3 (0.3) | 1.6 (0.4) | 1.8 (0.5) | 2.2 (0.6) |  | 1.7 (0.5)
  2 Year: number analyzed (Participants) | 8 | 42 | 64 | 48 | 17 | 0 | 179
  2 Year | 1.0 (0.4) | 1.3 (0.3) | 1.6 (0.4) | 1.9 (0.5) | 1.8 (0.5) |  | 1.6 (0.5)

9. Other Pre Specified Outcome: Subject's Average Effective Orifice Area Measurements - 11000M
Description: Effective orifice area represents the cross-sectional area of the blood flow downstream of the mitral valve. Effective orifice area is evaluated by echocardiography over time.
Time Frame: 3 Months, 1 Year, and 2 Years Post Implant
Population: The outcome is reported for subjects who received the Model 11000M device where data is available.
Measure: Mean (Standard Deviation); unit: Centimeters Squared
Arm/Group | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 25mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 27mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 29mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 31mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 33mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - Total
Number analyzed (Participants) | 6 | 29 | 25 | 16 | 6 | 82
Centimeters Squared
  3 Months: number analyzed (Participants) | 5 | 26 | 20 | 14 | 6 | 71
  3 Months | 1.2 (0.3) | 1.4 (0.4) | 1.6 (0.6) | 1.6 (0.4) | 1.8 (0.4) | 1.5 (0.5)
  1 Year: number analyzed (Participants) | 4 | 23 | 20 | 12 | 6 | 65
  1 Year | 1.1 (0.4) | 1.2 (0.3) | 1.5 (0.6) | 1.4 (0.5) | 1.5 (0.7) | 1.4 (0.5)
  2 Year: number analyzed (Participants) | 0 | 13 | 6 | 2 | 2 | 23
  2 Year |  | 1.3 (0.5) | 1.4 (0.4) | 1.6 (0.0) | 1.2 (0.3) | 1.4 (0.4)

10. Other Pre Specified Outcome: Subject's Average Effective Orifice Area Index (EOAI) Measurements - 11000A
Description: Effective orifice area index represents the minimal cross-sectional area of the blood flow downstream of the aortic valve divided by the person's body surface area. Effective orifice area index is evaluated by echocardiography over time.
Time Frame: 3 Months, 1 Year, and 2 Years Post Implant
Population: The outcome is reported for subjects who received the Model 11000A device where data is available.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 19mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 21mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 23mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 25mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 27mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 29mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - Total
Number analyzed (Participants) | 22 | 131 | 214 | 202 | 100 | 20 | 689
cm^2/m^2
  3 Months: number analyzed (Participants) | 22 | 117 | 196 | 184 | 90 | 11 | 620
  3 Months | 0.8 (0.3) | 0.8 (0.3) | 0.9 (0.3) | 0.9 (0.3) | 1.1 (0.3) | 1.1 (0.3) | 0.9 (0.3)
  1 Year: number analyzed (Participants) | 16 | 97 | 155 | 131 | 68 | 0 | 467
  1 Year | 0.6 (0.1) | 0.7 (0.2) | 0.8 (0.2) | 0.8 (0.2) | 1.0 (0.3) |  | 0.8 (0.3)
  2 Year: number analyzed (Participants) | 8 | 42 | 64 | 48 | 17 | 0 | 179
  2 Year | 0.6 (0.3) | 0.7 (0.2) | 0.8 (0.2) | 0.9 (0.2) | 0.8 (0.2) |  | 0.8 (0.2)

11. Other Pre Specified Outcome: Subject's Average Effective Orifice Area Index (EOAI) Measurements - 11000M
Description: Effective orifice area index represents the minimal cross-sectional area of the blood flow downstream of the mitral valve divided by the person's body surface area. Effective orifice area index is evaluated by echocardiography over time.
Time Frame: 3 Months, 1 Year, and 2 Years Post Implant
Population: The outcome is reported for subjects who received the Model 11000M device where data is available.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 25mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 27mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 29mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 31mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 33mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - Total
Number analyzed (Participants) | 6 | 29 | 25 | 16 | 6 | 82
cm^2/m^2
  3 Months: number analyzed (Participants) | 5 | 26 | 20 | 14 | 6 | 71
  3 Months | 0.7 (0.2) | 0.8 (0.3) | 0.8 (0.3) | 0.8 (0.2) | 0.9 (0.2) | 0.8 (0.3)
  1 Year: number analyzed (Participants) | 4 | 23 | 20 | 12 | 6 | 65
  1 Year | 0.6 (0.2) | 0.7 (0.2) | 0.8 (0.3) | 0.7 (0.2) | 0.7 (0.3) | 0.7 (0.2)
  2 Year: number analyzed (Participants) | 0 | 13 | 6 | 2 | 2 | 23
  2 Year |  | 0.8 (0.3) | 0.7 (0.2) | 0.9 (0.2) | 0.6 (0.1) | 0.7 (0.3)

12. Other Pre Specified Outcome: Subject's Average Performance Index Measurements - 11000A
Description: Performance index is defined as the subject's effective orifice area (the cross sectional area of the blood flow downstream of the aortic valve) divided by the subject's native orifice area. Effective orifice area is evaluated by echocardiography over time.
Time Frame: 3 Months, 1 Year, and 2 Years Post Implant
Population: The outcome is reported for subjects who received the Model 11000A device where data is available.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 19mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 21mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 23mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 25mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 27mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 29mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - Total
Number analyzed (Participants) | 22 | 131 | 214 | 202 | 100 | 20 | 689
cm^2/m^2
  3 Months: number analyzed (Participants) | 22 | 117 | 196 | 184 | 90 | 11 | 620
  3 Months | 1.1 (0.3) | 0.9 (0.2) | 0.9 (0.2) | 0.9 (0.2) | 0.9 (0.3) | 0.8 (0.3) | 0.9 (0.2)
  1 Year: number analyzed (Participants) | 16 | 97 | 155 | 131 | 68 | 0 | 467
  1 Year | 0.9 (0.2) | 0.8 (0.2) | 0.8 (0.2) | 0.8 (0.2) | 0.9 (0.2) |  | 0.8 (0.2)
  2 Year: number analyzed (Participants) | 8 | 42 | 64 | 48 | 17 | 0 | 179
  2 Year | 0.8 (0.3) | 0.8 (0.2) | 0.8 (0.2) | 0.9 (0.2) | 0.7 (0.2) |  | 0.8 (0.2)

13. Other Pre Specified Outcome: Subject's Average Performance Index Measurements - 11000M
Description: Performance index is defined as the subject's effective orifice area (the crosssectional area of the blood flow downstream of the mitral valve) divided by the subject's native orifice area. Effective orifice area is evaluated by echocardiography over time.
Time Frame: 3 Months, 1 Year, and 2 Years Post Implant
Population: The outcome is reported for subjects who received the Model 11000M device where data is available.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 25mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 27mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 29mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 31mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 33mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - Total
Number analyzed (Participants) | 6 | 29 | 25 | 16 | 6 | 82
cm^2/m^2
  3 Months: number analyzed (Participants) | 5 | 26 | 21 | 14 | 6 | 72
  3 Months | 0.6 (0.2) | 0.6 (0.2) | 0.6 (0.2) | 0.5 (0.1) | 0.6 (0.1) | 0.6 (0.2)
  1 Year: number analyzed (Participants) | 4 | 23 | 20 | 13 | 6 | 66
  1 Year | 0.6 (0.2) | 0.6 (0.2) | 0.6 (0.2) | 0.5 (0.2) | 0.5 (0.2) | 0.5 (0.2)
  2 Year: number analyzed (Participants) | 0 | 13 | 6 | 2 | 2 | 23
  2 Year |  | 0.6 (0.2) | 0.6 (0.2) | 0.6 (0.0) | 0.4 (0.1) | 0.6 (0.2)

14. Other Pre Specified Outcome: Subject's Average Cardiac Output Over Time - 11000A
Description: The amount of blood the heart pumps through the circulatory system in a minute.
Time Frame: 3 Months, 1 Year, and 2 Years Post Implant
Population: The outcome is reported for subjects who received the Model 11000A device where data is available.
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 19mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 21mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 23mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 25mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 27mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 29mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - Total
Number analyzed (Participants) | 22 | 131 | 214 | 202 | 100 | 20 | 689
Liters/minute
  3 Months: number analyzed (Participants) | 22 | 118 | 196 | 184 | 90 | 11 | 621
  3 Months | 5.1 (1.3) | 4.5 (1.2) | 4.7 (1.4) | 4.8 (1.2) | 5.2 (1.8) | 4.4 (1.2) | 4.8 (1.4)
  1 Year: number analyzed (Participants) | 16 | 97 | 156 | 131 | 68 | 0 | 468
  1 Year | 4.5 (0.9) | 4.7 (1.8) | 4.4 (1.2) | 4.8 (1.7) | 5.4 (1.6) |  | 4.7 (1.6)
  2 Year: number analyzed (Participants) | 8 | 42 | 64 | 47 | 18 | 0 | 179
  2 Year | 3.7 (1.1) | 4.3 (1.1) | 4.4 (1.2) | 4.9 (1.7) | 4.4 (1.4) |  | 4.5 (1.4)

15. Other Pre Specified Outcome: Subject's Average Cardiac Output Over Time - 11000M
Description: The amount of blood the heart pumps through the circulatory system in a minute.
Time Frame: 3 Months, 1 Year, and 2 Years Post Implant
Population: The outcome is reported for subjects who received the Model 11000M device where data is available.
Measure: Mean (Standard Deviation); unit: Liters/Minute
Arm/Group | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 25mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 27mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 29mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 31mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 33mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - Total
Number analyzed (Participants) | 6 | 29 | 25 | 16 | 6 | 82
Liters/Minute
  3 Months: number analyzed (Participants) | 5 | 26 | 21 | 15 | 6 | 73
  3 Months | 4.0 (1.2) | 3.6 (0.9) | 4.3 (1.4) | 3.9 (0.8) | 4.6 (1.0) | 4.0 (1.1)
  1 Year: number analyzed (Participants) | 4 | 23 | 21 | 13 | 6 | 67
  1 Year | 3.7 (1.0) | 3.3 (1.1) | 4.4 (1.9) | 3.8 (1.1) | 3.8 (0.8) | 3.8 (1.4)
  2 Year: number analyzed (Participants) | 0 | 13 | 7 | 2 | 2 | 24
  2 Year |  | 3.3 (1.1) | 4.1 (1.3) | 3.6 (0.3) | 3.3 (0.6) | 3.6 (1.1)

16. Other Pre Specified Outcome: Subject's Average Cardiac Index Over Time- 11000A
Description: Cardiac index is an assessment that divides the cardiac output from left ventricle in one minute by the person's body surface area (BSA), thus relating heart performance to the size of the individual.
Time Frame: 3 Months, 1 Year, and 2 Years Post Implant
Population: The outcome is reported for subjects who received the Model 11000A device where data is available.
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 19mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 21mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 23mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 25mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 27mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 29mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - Total
Number analyzed (Participants) | 22 | 131 | 214 | 202 | 100 | 20 | 689
L/min/m^2
  3 Months: number analyzed (Participants) | 22 | 118 | 196 | 184 | 90 | 11 | 621
  3 Months | 3.0 (0.8) | 2.4 (0.7) | 2.4 (0.8) | 2.3 (0.6) | 2.4 (0.9) | 2.0 (0.4) | 2.4 (0.7)
  1 Year: number analyzed (Participants) | 16 | 97 | 156 | 131 | 67 | 0 | 467
  1 Year | 2.6 (0.5) | 2.5 (1.0) | 2.2 (0.6) | 2.2 (0.8) | 2.4 (0.7) |  | 2.3 (0.8)
  2 Year: number analyzed (Participants) | 8 | 42 | 64 | 47 | 18 | 0 | 179
  2 Year | 2.2 (0.8) | 2.3 (0.6) | 2.2 (0.7) | 2.3 (0.7) | 2.0 (0.6) |  | 2.2 (0.7)

17. Other Pre Specified Outcome: Subject's Average Cardiac Index Over Time - 11000M
Description: Cardiac index is an assessment that divides the cardiac output from left ventricle in one minute by the person's body surface area(BSA), thus relating heart performance to the size of the individual.
Time Frame: 3 Months, 1 Year, and 2 Years Post Implant
Population: The outcome is reported for subjects who received the Model 11000M device where data is available.
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 25mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 27mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 29mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 31mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 33mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - Total
Number analyzed (Participants) | 6 | 29 | 25 | 16 | 6 | 82
L/min/m^2
  3 Months: number analyzed (Participants) | 5 | 26 | 21 | 15 | 6 | 73
  3 Months | 2.2 (0.7) | 2.1 (0.6) | 2.2 (0.6) | 1.9 (0.4) | 2.1 (0.8) | 2.1 (0.6)
  1 Year: number analyzed (Participants) | 4 | 23 | 21 | 13 | 6 | 67
  1 Year | 2.0 (0.5) | 1.9 (0.5) | 2.2 (0.9) | 1.9 (0.5) | 1.8 (0.4) | 2.0 (0.7)
  2 Year: number analyzed (Participants) | 0 | 13 | 7 | 2 | 2 | 24
  2 Year |  | 1.9 (0.7) | 2.1 (0.5) | 1.9 (0.3) | 1.6 (0.3) | 1.9 (0.6)

18. Other Pre Specified Outcome: Subject's Amount of Total Valvular Regurgitation Over Time - 11000A
Description: Valvular regurgitation occurs when the valve in the heart does not close tightly allowing some of the blood that was pumped out of the heart to leak back into it. Valvular regurgitation is evaluated by echocardiography over time. It is assessed on a scale from 0 to 4, where 0 represents no regurgitation and 4 represents severe regurgitation.
Time Frame: 3 Months, 1 Year, and 2 Years Post Implant
Population: The outcome is reported for subjects who received the Model 11000A device where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 19mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 21mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 23mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 25mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 27mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 29mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - Total
Number analyzed (Participants) | 22 | 131 | 214 | 202 | 100 | 20 | 689
Participants
  3 Months: number analyzed (Participants) | 21 | 118 | 196 | 186 | 90 | 12 | 623
  3 Months: 0 None | 17 | 106 | 166 | 162 | 69 | 11 | 531
  3 Months: +1 Trivial/Trace | 3 | 11 | 25 | 20 | 20 | 1 | 80
  3 Months: +2 Mild | 1 | 1 | 3 | 4 | 1 | 0 | 10
  3 Months: +3 Moderate | 0 | 0 | 1 | 0 | 0 | 0 | 1
  3 Months: +4 Severe | 0 | 0 | 1 | 0 | 0 | 0 | 1
  1 Year: number analyzed (Participants) | 16 | 97 | 159 | 131 | 68 | 0 | 471
  1 Year: 0 None | 11 | 88 | 125 | 112 | 49 |  | 385
  1 Year: +1 Trivial/Trace | 3 | 6 | 26 | 12 | 17 |  | 64
  1 Year: +2 Mild | 2 | 2 | 8 | 7 | 2 |  | 21
  1 Year: +3 Moderate | 0 | 1 | 0 | 0 | 0 |  | 1
  1 Year: +4 Severe | 0 | 0 | 0 | 0 | 0 |  | 0
  2 Year: number analyzed (Participants) | 8 | 42 | 66 | 49 | 18 | 0 | 183
  2 Year: 0 None | 4 | 32 | 51 | 38 | 11 |  | 136
  2 Year: +1 Trivial/Trace | 2 | 5 | 11 | 9 | 5 |  | 32
  2 Year: +2 Mild | 2 | 5 | 3 | 2 | 2 |  | 14
  2 Year: +3 Moderate | 0 | 0 | 1 | 0 | 0 |  | 1
  2 Year: +4 Severe | 0 | 0 | 0 | 0 | 0 |  | 0

19. Other Pre Specified Outcome: Subject's Amount of Total Valvular Regurgitation Over Time - 11000M
Description: Mitral valvular regurgitation occurs when the mitral valve in the heart does not close tightly allowing some of the blood that was pumped out of the heart to leak back into it. Mitral valvular regurgitation is evaluated by echocardiography over time. It is assessed on a scale from 0 to 4, where 0 represents no regurgitation and 4 represents severe regurgitation.
Time Frame: 3 Months, 1 Year, and 2 Years Post Implant
Population: The outcome is reported for subjects who received the Model 11000M device where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 25mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 27mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 29mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 31mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 33mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - Total
Number analyzed (Participants) | 6 | 29 | 25 | 16 | 6 | 82
Participants
  3 Months: number analyzed (Participants) | 5 | 26 | 23 | 15 | 6 | 75
  3 Months: 0 None | 4 | 15 | 18 | 10 | 4 | 51
  3 Months: +1 Trivial/Trace | 1 | 7 | 5 | 3 | 2 | 18
  3 Months: +2 Mild | 0 | 3 | 0 | 2 | 0 | 5
  3 Months: +3 Moderate | 0 | 1 | 0 | 0 | 0 | 1
  3 Months: +4 Severe | 0 | 0 | 0 | 0 | 0 | 0
  1 Year: number analyzed (Participants) | 4 | 25 | 21 | 13 | 6 | 69
  1 Year: 0 None | 3 | 15 | 13 | 8 | 3 | 42
  1 Year: +1 Trivial/Trace | 1 | 5 | 7 | 4 | 2 | 19
  1 Year: +2 Mild | 0 | 4 | 0 | 0 | 1 | 5
  1 Year: +3 Moderate | 0 | 1 | 1 | 0 | 0 | 2
  1 Year: +4 Severe | 0 | 0 | 0 | 1 | 0 | 1
  2 Year: number analyzed (Participants) | 0 | 13 | 7 | 2 | 2 | 24
  2 Year: 0 None |  | 6 | 6 | 1 | 0 | 13
  2 Year: +1 Trivial/Trace |  | 2 | 1 | 1 | 2 | 6
  2 Year: +2 Mild |  | 4 | 0 | 0 | 0 | 4
  2 Year: +3 Moderate |  | 1 | 0 | 0 | 0 | 1
  2 Year: +4 Severe |  | 0 | 0 | 0 | 0 | 0

20. Other Pre Specified Outcome: Subject's Amount of Paravalvular Leak Over Time - 11000A
Description: Paravalvular leak refers to blood flowing through a channel between the implanted artificial valve and the cardiac tissue as a result of inappropriate sealing.
  Paravalvular leak is evaluated by echocardiography over time. It is assessed on a scale from minimum of 0 to maximum of 4, where 0 = no leak, 1 = a trace leak, 2 = a mild leak, 3 = a moderate leak, and 4 = a severe leak. Higher numbers on the scale show a worsening outcome.
Time Frame: 3 Months, 1 Year, and 2 Years Post Implant
Population: The outcome is reported for subjects who received the Model 11000A device where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 19mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 21mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 23mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 25mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 27mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - 29mm | Edwards Pericardial Aortic Bioprosthesis, Model 11000A - Total
Number analyzed (Participants) | 22 | 131 | 214 | 202 | 100 | 20 | 689
Participants
  3 Months: number analyzed (Participants) | 21 | 118 | 195 | 185 | 90 | 12 | 621
  3 Months: 0 None | 20 | 118 | 191 | 182 | 87 | 12 | 610
  3 Months: +1 Trivial/Trace | 1 | 0 | 3 | 1 | 2 | 0 | 7
  3 Months: +2 Mild | 0 | 0 | 0 | 2 | 1 | 0 | 3
  3 Months: +3 Moderate | 0 | 0 | 1 | 0 | 0 | 0 | 1
  3 Months: +4 Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  1 Year: number analyzed (Participants) | 15 | 96 | 158 | 130 | 69 | 0 | 468
  1 Year: 0 None | 12 | 92 | 152 | 127 | 67 |  | 450
  1 Year: +1 Trivial/Trace | 2 | 1 | 3 | 2 | 0 |  | 8
  1 Year: +2 Mild | 1 | 3 | 3 | 1 | 2 |  | 10
  1 Year: +3 Moderate | 0 | 0 | 0 | 0 | 0 |  | 0
  1 Year: +4 Severe | 0 | 0 | 0 | 0 | 0 |  | 0
  2 Year: number analyzed (Participants) | 8 | 42 | 66 | 48 | 18 | 0 | 182
  2 Year: 0 None | 6 | 37 | 61 | 46 | 16 |  | 166
  2 Year: +1 Trivial/Trace | 0 | 1 | 2 | 1 | 2 |  | 6
  2 Year: +2 Mild | 2 | 4 | 2 | 1 | 0 |  | 9
  2 Year: +3 Moderate | 0 | 0 | 1 | 0 | 0 |  | 1
  2 Year: +4 Severe | 0 | 0 | 0 | 0 | 0 |  | 0

21. Other Pre Specified Outcome: Subject's Amount of Paravalvular Leak Over Time - 11000M
Description: as for outcome 20
Time Frame: 3 Months, 1 Year, and 2 Years Post Implant
Population: The outcome is reported for subjects who received the Model 11000M device where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 25mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 27mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 29mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 31mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - 33mm | Edwards Pericardial Mitral Bioprosthesis, Model 11000M - Total
Number analyzed (Participants) | 6 | 29 | 25 | 16 | 6 | 82
Participants
  3 Months: number analyzed (Participants) | 5 | 26 | 23 | 15 | 6 | 75
  3 Months: 0 None | 5 | 26 | 23 | 15 | 6 | 75
  3 Months: +1 Trivial/Trace | 0 | 0 | 0 | 0 | 0 | 0
  3 Months: +2 Mild | 0 | 0 | 0 | 0 | 0 | 0
  3 Months: +3 Moderate | 0 | 0 | 0 | 0 | 0 | 0
  3 Months: +4 Severe | 0 | 0 | 0 | 0 | 0 | 0
  1 Year: number analyzed (Participants) | 4 | 25 | 21 | 13 | 6 | 69
  1 Year: 0 None | 4 | 25 | 21 | 11 | 6 | 67
  1 Year: +1 Trivial/Trace | 0 | 0 | 0 | 2 | 0 | 2
  1 Year: +2 Mild | 0 | 0 | 0 | 0 | 0 | 0
  1 Year: +3 Moderate | 0 | 0 | 0 | 0 | 0 | 0
  1 Year: +4 Severe | 0 | 0 | 0 | 0 | 0 | 0
  2 Year: number analyzed (Participants) | 0 | 13 | 7 | 2 | 2 | 24
  2 Year: 0 None |  | 13 | 7 | 2 | 2 | 24
  2 Year: +1 Trivial/Trace |  | 0 | 0 | 0 | 0 | 0
  2 Year: +2 Mild |  | 0 | 0 | 0 | 0 | 0
  2 Year: +3 Moderate |  | 0 | 0 | 0 | 0 | 0
  2 Year: +4 Severe |  | 0 | 0 | 0 | 0 | 0

22. Other Pre Specified Outcome: Subject's New York Heart Association (NYHA) Functional Class Compared to Baseline
Description: The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life.
  Class I. No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  Class II. Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  Class III. Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV. Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
Time Frame: 3 Months, 1 Year, and 2 Years Post Implant
Population: The outcome is reported for subjects who received the Model 11000A or Model 11000M device where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A | Edwards Pericardial Mitral Bioprosthesis, Model 11000M
Number analyzed (Participants) | 689 | 82
Participants
  3 Months: number analyzed (Participants) | 645 | 75
  3 Months: Improved | 431 | 66
  3 Months: Same | 200 | 7
  3 Months: Worsened | 14 | 2
  1 Year: number analyzed (Participants) | 509 | 73
  1 Year: Improved | 331 | 66
  1 Year: Same | 161 | 7
  1 Year: Worsened | 17 | 0
  2 Year: number analyzed (Participants) | 240 | 29
  2 Year: Improved | 157 | 26
  2 Year: Same | 75 | 3
  2 Year: Worsened | 8 | 0

23. Other Pre Specified Outcome: Subject's Average Score at Baseline and 1 Year on the Quality of Life Survey
Description: The Medical Outcomes Study Short-Form 12 (SF-12) contains two components - the Physical Component Summary (PCS) and the Mental Component Summary (MCS).
  The SF-12 Physical Component Summary questionnaire scale ranges from a maximum of 100, which reflects the best health status to a minimum of 0, which reflects the worst health status.
  The SF-12 Mental Component Summary scale ranges from a maximum of 100, which reflects the best health status to a minimum of 0, which reflects the worst health status.
Time Frame: Baseline and one year post-implant
Population: The outcome is reported for subjects who received the Model 11000A or Model 11000M device where data is available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A | Edwards Pericardial Mitral Bioprosthesis, Model 11000M
Number analyzed (Participants) | 689 | 82
units on a scale
  Physical Health-Baseline: number analyzed (Participants) | 485 | 71
  Physical Health-Baseline | 42.9 (9.7) | 40.1 (8.9)
  Physical Health-1 Year: number analyzed (Participants) | 485 | 71
  Physical Health-1 Year | 49.1 (9.2) | 48.8 (7.0)
  Mental Health-Baseline: number analyzed (Participants) | 485 | 71
  Mental Health-Baseline | 50.9 (9.5) | 49.2 (11.5)
  Mental Health-1 Year: number analyzed (Participants) | 485 | 71
  Mental Health-1 Year | 53.8 (8.5) | 52.3 (9.3)

24. Other Pre Specified Outcome: Subject's Average White Blood Cell Count
Description: Laboratory analysis of White Blood Cell (WBC) count on blood drawn from subject; WBC fight infection.
Time Frame: Baseline, Discharge, 3 Months, 1 Year and 2 Year
Population: The outcome is reported for subjects who received the Model 11000A or Model 11000M device where data is available.
Measure: Mean (Standard Deviation); unit: 10^3 cells /microliter
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A | Edwards Pericardial Mitral Bioprosthesis, Model 11000M
Number analyzed (Participants) | 689 | 82
10^3 cells /microliter
  Baseline | 7.2 (1.9) | 7.4 (2.6)
  Discharge: number analyzed (Participants) | 682 | 82
  Discharge | 9.1 (2.8) | 10.4 (5.3)
  3 Months: number analyzed (Participants) | 621 | 75
  3 Months | 7.1 (1.7) | 7.1 (2.0)
  1 Year: number analyzed (Participants) | 499 | 72
  1 Year | 7.3 (1.9) | 7.1 (2.3)
  2 Year: number analyzed (Participants) | 225 | 30
  2 Year | 7.3 (1.8) | 7.4 (1.8)

25. Other Pre Specified Outcome: Subject's Average Red Blood Cells Count
Description: Laboratory Analysis of Red Blood Cell (RBC) Count on blood drawn from subjects; RBC carry oxygen.
Time Frame: Baseline, Discharge, 3 Months, 1 Year and 2 Year
Population: The outcome is reported for subjects who received the Model 11000A or Model 11000M device where data is available.
Measure: Mean (Standard Deviation); unit: 10^6 cells/microliters
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A | Edwards Pericardial Mitral Bioprosthesis, Model 11000M
Number analyzed (Participants) | 689 | 82
10^6 cells/microliters
  Baseline | 4.5 (0.5) | 4.4 (0.6)
  Discharge: number analyzed (Participants) | 682 | 82
  Discharge | 3.3 (0.5) | 3.3 (0.4)
  3 Months: number analyzed (Participants) | 621 | 75
  3 Months | 4.7 (0.5) | 4.5 (0.7)
  1 Year: number analyzed (Participants) | 498 | 72
  1 Year | 4.7 (0.5) | 4.5 (0.6)
  2 Year: number analyzed (Participants) | 225 | 30
  2 Year | 4.6 (0.5) | 4.6 (0.5)

26. Other Pre Specified Outcome: Subject's Average Hematocrit Percentage
Description: Laboratory Analysis of Hematocrit Percentage on blood drawn from subjects. Hematocrit is the proportion of red blood cells to the plasma (liquid portion of the blood).
Time Frame: Baseline, Discharge, 3 Months, 1 Year and 2 Year
Population: The outcome is reported for subjects who received the Model 11000A or 11000M device where data is available.
Measure: Mean (Standard Deviation); unit: percentage of red blood cells
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A | Edwards Pericardial Mitral Bioprosthesis, Model 11000M
Number analyzed (Participants) | 689 | 82
percentage of red blood cells
  Baseline | 41.0 (4.0) | 40.3 (4.6)
  Discharge: number analyzed (Participants) | 682 | 82
  Discharge | 30.1 (4.1) | 30.1 (3.9)
  3 Months: number analyzed (Participants) | 621 | 75
  3 Months | 41.0 (4.2) | 39.3 (5.3)
  1 Year: number analyzed (Participants) | 499 | 72
  1 Year | 41.9 (4.1) | 41.3 (4.8)
  2 Year: number analyzed (Participants) | 225 | 30
  2 Year | 42.0 (3.9) | 42.4 (4.3)

27. Other Pre Specified Outcome: Subject's Average Hemoglobin Count
Description: Laboratory Analysis of Hemoglobin Count on blood drawn from subjects. Hemoglobin is an oxygen-carrying protein in red blood cells.
Time Frame: Baseline, Discharge, 3 Months, 1 Year and 2 Year
Population: The outcome is reported for subjects who received the Model 11000A or 11000M device where data is available.
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A | Edwards Pericardial Mitral Bioprosthesis, Model 11000M
Number analyzed (Participants) | 689 | 82
g/dl
  Baseline | 13.8 (1.5) | 13.3 (1.6)
  Discharge: number analyzed (Participants) | 682 | 82
  Discharge | 10.0 (1.4) | 9.9 (1.2)
  3 Months: number analyzed (Participants) | 621 | 75
  3 Months | 13.5 (1.6) | 12.7 (1.9)
  1 Year: number analyzed (Participants) | 499 | 72
  1 Year | 14.0 (1.7) | 13.6 (1.6)
  2 Year: number analyzed (Participants) | 225 | 30
  2 Year | 14.0 (1.5) | 14.0 (1.3)

28. Other Pre Specified Outcome: Subject's Average Platelet Count
Description: Laboratory Analysis of Platelet Count on blood drawn from subjects; platelets help with blood clotting.
Time Frame: Baseline, Discharge, 3 Months, 1 Year, and 2 Years
Population: The outcome is reported for subjects who received the Model 11000A or 11000M device where data is available.
Measure: Mean (Standard Deviation); unit: 10^3 platelets per microliter
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A | Edwards Pericardial Mitral Bioprosthesis, Model 11000M
Number analyzed (Participants) | 689 | 82
10^3 platelets per microliter
  Baseline | 208.6 (59.0) | 203.6 (52.1)
  Discharge: number analyzed (Participants) | 682 | 82
  Discharge | 217.7 (90.1) | 196.0 (75.3)
  3 Months: number analyzed (Participants) | 621 | 75
  3 Months | 215.3 (62.6) | 221.0 (71.8)
  1 Year: number analyzed (Participants) | 499 | 72
  1 Year | 207.7 (65.8) | 207.8 (51.7)
  2 Year: number analyzed (Participants) | 225 | 30
  2 Year | 200.6 (54.5) | 204.0 (54.1)

29. Other Pre Specified Outcome: Subject's Average Plasma Free Hemoglobin
Description: Laboratory Analysis of Plasma Free Hemoglobin on blood drawn from subjects. This blood test measures the level of free hemoglobin in the plasma (liquid portion of the blood).
Time Frame: Baseline, Discharge, 3 Months, 1 Year and 2 Year
Population: The outcome is reported for subjects who received the Model 11000A or 11000M device where data is available.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A | Edwards Pericardial Mitral Bioprosthesis, Model 11000M
Number analyzed (Participants) | 689 | 82
mg/dl
  Baseline: number analyzed (Participants) | 629 | 63
  Baseline | 11.6 (18.4) | 19.8 (32.5)
  Discharge: number analyzed (Participants) | 560 | 54
  Discharge | 7.3 (12.2) | 7.2 (6.5)
  3 Months: number analyzed (Participants) | 582 | 56
  3 Months | 12.4 (22.2) | 10.6 (12.1)
  1 Year: number analyzed (Participants) | 463 | 48
  1 Year | 13.8 (25.5) | 8.6 (12.3)
  2 Year: number analyzed (Participants) | 216 | 16
  2 Year | 17.3 (33.9) | 20.5 (33.9)

30. Other Pre Specified Outcome: Subject's Average International Normalized Ratio
Description: Laboratory Analysis of International Normalized Ratio (INR) on blood drawn from subjects. The INR is a calculation based on results of a prothrombin time (PT). The PT is a blood test that measures the time it takes for the plasma (liquid portion of the blood) to clot. INR results will vary according to a person's age, the medicines they take, and any health problems they may have. In general, the higher the INR number, the longer it takes for the blood to clot. In healthy people an INR of 1.1 or below is considered normal. An INR range of 2.0 to 3.0 is generally an effective therapeutic range for people taking blood thinner medication.
Time Frame: Baseline, Discharge, 3 Months, 1 Year and 2 Year
Population: The outcome is reported for subjects who received the Model 11000A or 11000M device where data is available.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A | Edwards Pericardial Mitral Bioprosthesis, Model 11000M
Number analyzed (Participants) | 689 | 82
Ratio
  Baseline: number analyzed (Participants) | 672 | 80
  Baseline | 1.1 (0.2) | 1.4 (0.7)
  Discharge: number analyzed (Participants) | 579 | 80
  Discharge | 1.3 (0.4) | 1.7 (0.6)
  3 Months: number analyzed (Participants) | 479 | 62
  3 Months | 1.3 (0.7) | 1.9 (0.8)
  1 Year: number analyzed (Participants) | 364 | 61
  1 Year | 1.2 (0.5) | 1.7 (0.8)
  2 Year: number analyzed (Participants) | 194 | 26
  2 Year | 1.2 (0.6) | 1.6 (0.8)

31. Other Pre Specified Outcome: Subject's Average Partial Thromboplastin Time
Description: Laboratory Analysis of partial thromboplastin time (PTT) on blood drawn from subjects. PTT is a blood test that looks at how long it takes for the blood to clot.
Time Frame: Baseline, Discharge, 3 Months, 1 Year and 2 Year
Population: The outcome is reported for subjects who received the Model 11000A or 11000M device where data is available.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A | Edwards Pericardial Mitral Bioprosthesis, Model 11000M
Number analyzed (Participants) | 689 | 82
Seconds
  Baseline: number analyzed (Participants) | 608 | 74
  Baseline | 30.0 (6.0) | 35.1 (14.4)
  Discharge: number analyzed (Participants) | 489 | 58
  Discharge | 32.1 (8.5) | 37.2 (14.5)
  3 Months: number analyzed (Participants) | 399 | 45
  3 Months | 31.2 (15.8) | 36.0 (8.1)
  1 Year: number analyzed (Participants) | 304 | 48
  1 Year | 29.4 (5.7) | 35.3 (14.3)
  2 Year: number analyzed (Participants) | 167 | 18
  2 Year | 31.4 (14.4) | 33.7 (9.5)

32. Other Pre Specified Outcome: Subject's Average Prothrombin Time
Description: Laboratory Analysis of Prothrombin Time (PT) on blood drawn from subjects. The PT is a blood test that measures the time it takes for the plasma (liquid portion of the blood) to clot.
Time Frame: Baseline, Discharge, 3 Months, 1 Year, and 2 Years
Population: The outcome is reported for subjects who received the Model 11000A or 11000M device where data is available.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A | Edwards Pericardial Mitral Bioprosthesis, Model 11000M
Number analyzed (Participants) | 689 | 82
Seconds
  Baseline: number analyzed (Participants) | 664 | 73
  Baseline | 12.7 (2.5) | 16.2 (8.0)
  Discharge: number analyzed (Participants) | 577 | 72
  Discharge | 15.0 (5.0) | 20.1 (7.3)
  3 Months: number analyzed (Participants) | 475 | 56
  3 Months | 15.2 (7.4) | 21.0 (8.4)
  1 Year: number analyzed (Participants) | 364 | 58
  1 Year | 13.8 (5.7) | 19.1 (8.8)
  2 Year: number analyzed (Participants) | 193 | 25
  2 Year | 14.1 (6.4) | 17.3 (7.9)

33. Other Pre Specified Outcome: Subjects Average Serum Glycerol Levels
Description: Laboratory analysis of serum glycerol in blood drawn from subjects. This blood test measures the amount of glycerol (a naturally occurring carbohydrate, that can be used as a fuel source by the body) in the serum (liquid portion of the blood).
Time Frame: Pre-Implant (post-heparinization) and Post-Implant (between 60 and 120 minutes after heart was restarted)
Population: The outcome is reported for subjects who received the Model 11000A device where data is available.
Measure: Mean (Standard Deviation); unit: micromol/L
Groups:
- Edwards Pericardial Bioprosthesis, Model 11000A: The Edwards Pericardial Aortic Bioprosthesis, Model 11000A, is indicated for patients who require replacement of their native or prosthetic aortic valve.
Arm/Group | Edwards Pericardial Bioprosthesis, Model 11000A
Number analyzed (Participants) | 689
micromol/L
  Pre-Implant: number analyzed (Participants) | 119
  Pre-Implant | 405.4 (270.2)
  Post-Implant: number analyzed (Participants) | 117
  Post-Implant | 245.6 (345.8)

ADVERSE EVENTS:
Time Frame: Events occurring from baseline through three years post implant for the 11000A, and four years post implant for 11000M.
Description: Adverse event table is reported for Subjects who received the Model 11000A or 11000M Device.
Arm/Group | Edwards Pericardial Aortic Bioprosthesis, Model 11000A | Edwards Pericardial Mitral Bioprosthesis, Model 11000M
All-Cause Mortality (participants affected / at risk) | 26/689 | 8/82
Serious Adverse Events (participants affected / at risk) | 317/689 | 58/82
Other Adverse Events (participants affected / at risk) | 542/589 | 66/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edwards Pericardial Aortic Bioprosthesis, Model 11000A (N=689) | Edwards Pericardial Mitral Bioprosthesis, Model 11000M (N=82)
Anemia - Bleeding related - Major (Blood and lymphatic system disorders) | 12 (12) | 2 (2)
Anemia - Bleeding related - Minor (Blood and lymphatic system disorders) | 11 (11) | 1 (1)
Anemia - Non-bleeding related (Blood and lymphatic system disorders) | 6 (6) | 3 (3)
Angina, stable (Cardiac disorders) | 1 (1) | 2 (2)
Angina, unstable (Cardiac disorders) | 3 (3) | 0 (0)
Arrhythmia - Atrial flutter (Cardiac disorders) | 7 (7) | 3 (3)
Arrhythmia - AV block - 1st degree (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia - AV block - 2nd degree (Cardiac disorders) | 4 (4) | 0 (0)
Arrhythmia - AV block - 3rd degree (Cardiac disorders) | 24 (24) | 6 (6)
Arrhythmia - Bradycardia (Cardiac disorders) | 4 (4) | 1 (1)
Arrhythmia - Bundle branch block - Left (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia - Bundle branch block - Right (Cardiac disorders) | 2 (2) | 0 (0)
Arrhythmia - Other (Cardiac disorders) | 10 (10) | 5 (5)
Arrhythmia - Paroxysmal Atrial Fibrillation (PAF) (Cardiac disorders) | 39 (41) | 8 (9)
Arrhythmia - Permanent atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Arrhythmia - Persistent atrial fibrillation (Cardiac disorders) | 14 (14) | 6 (6)
Arrhythmia - Supraventricular Tachycardia (SVT) (Cardiac disorders) | 3 (3) | 1 (1)
Arrhythmia - Tachy-bradycardia (Cardiac disorders) | 4 (4) | 1 (1)
Arrhythmia - Tachycardia - Ventricular (Cardiac disorders) | 2 (2) | 0 (0)
Arrhythmia - Ventricular fibrillation (Cardiac disorders) | 4 (4) | 0 (0)
Biliary (gallbladder) (Gastrointestinal disorders) | 5 (6) | 1 (2)
Bleeding - Cardiovascular - Major (Blood and lymphatic system disorders) | 21 (21) | 3 (3)
Bleeding - Cardiovascular - Minor (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
Bleeding - Gastrointestinal lower - Major (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Bleeding - Gastrointestinal lower - Minor (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bleeding - Gastrointestinal upper - Major (Blood and lymphatic system disorders) | 4 (5) | 2 (2)
Bleeding - Genitourinary - Minor (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bleeding - Musculoskeletal/Dermatological - Major (e.g. ecchymosis) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bleeding - Neurological - Minor (e.g. CVA) (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Bleeding - Peripheral vascular - Minor (e.g. nosebleeds; hematomas) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bleeding - Pulmonary/Respiratory - Major (e.g. hemothorax) (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Blood sepsis (Blood and lymphatic system disorders) | 9 (10) | 3 (4)
Blood/Lymphatic - Other (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Bone fracture/Break (Musculoskeletal and connective tissue disorders) | 8 (9) | 1 (1)
Cancer - Newly diagnosed (General disorders) | 9 (9) | 1 (1)
Cancer - Progression of underlying disease (General disorders) | 4 (4) | 0 (0)
Cardiac arrest (Cardiac disorders) | 6 (6) | 3 (3)
Cardiac decompensation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 6 (6) | 1 (1)
Cardiovascular - Other (Cardiac disorders) | 23 (24) | 6 (7)
Coronary artery ostial obstruction (Cardiac disorders) | 2 (2) | 0 (0)
Endocarditis (Cardiac disorders) | 7 (7) | 2 (2)
Endocrine complications (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever - Unknown origin (General disorders) | 1 (1) | 0 (0)
Gastrointestinal - Esophageal rupture/tear (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal - Infection (Gastrointestinal disorders) | 7 (8) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 20 (25) | 2 (2)
Genitourinary - Other (Renal and urinary disorders) | 9 (10) | 1 (1)
Heart failure - Acute (Cardiac disorders) | 7 (7) | 5 (5)
Heart Failure - Chronic (CHF) (Cardiac disorders) | 11 (13) | 3 (7)
Hepatic complication - Other (Gastrointestinal disorders) | 3 (3) | 0 (0)
Hypertension - Systemic (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 8 (8) | 4 (4)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Infection/Inflammation - Other (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Metabolic complications (Gastrointestinal disorders) | 2 (2) | 0 (0)
Muscular skeletal/Dermatologic - Other (Musculoskeletal and connective tissue disorders) | 27 (31) | 5 (5)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Nonspecific, unknown, or other body system - Other complication (General disorders) | 43 (51) | 4 (4)
NSD - Paravalvular leak +2 Minor (General disorders) | 0 (0) | 1 (1)
NSD - Paravalvular leak +3 Major (General disorders) | 1 (1) | 1 (1)
NSD - Paravalvular leak +4 Major (General disorders) | 1 (1) | 0 (0)
Pancreatic complication (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pericardial effusion - Major (Cardiac disorders) | 8 (9) | 2 (2)
Pericardial effusion - Minor (Cardiac disorders) | 6 (6) | 0 (0)
Pericardial tamponade (Cardiac disorders) | 10 (10) | 1 (1)
Pericarditis (Cardiac disorders) | 5 (6) | 0 (0)
Pleural effusion - Bilateral (Cardiac disorders) | 13 (13) | 1 (1)
Pleural effusion - Left (Cardiac disorders) | 7 (9) | 3 (3)
Pleural effusion - Right (Cardiac disorders) | 15 (15) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 1 (1)
Psychiatric - Other (Psychiatric disorders) | 7 (7) | 1 (1)
Psychiatric disorder (Psychiatric disorders) | 1 (3) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism - Bilateral (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary/Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0)
Regurgitation - Tricuspid-indeterminate +4 (Cardiac disorders) | 0 (0) | 1 (2)
Renal dysfunction (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal - Other (Renal and urinary disorders) | 5 (6) | 0 (0)
Renal failure - Acute (Renal and urinary disorders) | 8 (9) | 5 (5)
Renal failure - Chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory dysfunction/Insufficiency (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 1 (1)
Respiratory failure - Acute Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Respiratory failure - COPD (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
Respiratory failure - Hemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure - Other (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 4 (4)
Respiratory failure - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Respiratory failure - Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Respiratory infection - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Respiratory infection - Upper (URI) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Speech disorder (General disorders) | 2 (2) | 0 (0)
Splenic complication (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sternal wound/Thoracic infection (Musculoskeletal and connective tissue disorders) | 13 (14) | 1 (1)
SVD - Study valve leaflet tear (General disorders) | 0 (0) | 1 (1)
Thrombocytopenia - Heparin Induced (HIT) (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia - Non-heparin induced (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thromboembolic event - Other - Central - No paresis (Cardiac disorders) | 0 (0) | 1 (1)
Thromboembolic event - Other - Peripheral - No paresis (Cardiac disorders) | 0 (0) | 1 (1)
Thromboembolic event - Stroke (Cardiac disorders) | 15 (17) | 3 (3)
Thromboembolic event - Transient Ischemic Attack (TIA) (Cardiac disorders) | 7 (9) | 0 (0)
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 4 (4) | 1 (1)
Valve thrombosis - Aortic (Cardiac disorders) | 0 (0) | 1 (1)
Vascular - Deep Vein Thrombosis (DVT) (Vascular disorders) | 3 (3) | 1 (1)
Vascular - Other (Vascular disorders) | 7 (9) | 0 (0)
Vision disorder (General disorders) | 1 (1) | 0 (0)
Wound infection - Other (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edwards Pericardial Aortic Bioprosthesis, Model 11000A (N=589) | Edwards Pericardial Mitral Bioprosthesis, Model 11000M (N=82)
Allergic reaction - Medication related (General disorders) | 4 (4) | 0 (0)
Allergic reaction - Other (General disorders) | 0 (0) | 1 (1)
Anemia - Bleeding related - Major (Blood and lymphatic system disorders) | 11 (11) | 2 (2)
Anemia - Bleeding related - Minor (Blood and lymphatic system disorders) | 87 (87) | 18 (18)
Anemia - Non-bleeding related (Blood and lymphatic system disorders) | 61 (61) | 14 (14)
Angina, stable (Cardiac disorders) | 5 (5) | 2 (2)
Angina, unstable (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia - Atrial flutter (Cardiac disorders) | 10 (10) | 5 (5)
Arrhythmia - AV block - 1st degree (Cardiac disorders) | 39 (40) | 11 (11)
Arrhythmia - AV block - 2nd degree (Cardiac disorders) | 7 (7) | 4 (4)
Arrhythmia - AV block - 3rd degree (Cardiac disorders) | 7 (7) | 2 (2)
Arrhythmia - Bradycardia (Cardiac disorders) | 17 (19) | 4 (4)
Arrhythmia - Bundle branch block - Left (Cardiac disorders) | 25 (25) | 0 (0)
Arrhythmia - Bundle branch block - Right (Cardiac disorders) | 28 (30) | 3 (3)
Arrhythmia - Other (Cardiac disorders) | 50 (50) | 8 (8)
Arrhythmia - Pacemaker/ICD malfunction (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia - Paroxysmal Atrial Fibrillation (PAF) (Cardiac disorders) | 136 (137) | 12 (12)
Arrhythmia - Paroxysmal Atrial Tachycardia (PAT) (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia - Permanent atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia - Persistent atrial fibrillation (Cardiac disorders) | 23 (23) | 3 (3)
Arrhythmia - Supraventricular Tachycardia (SVT) (Cardiac disorders) | 4 (4) | 1 (1)
Arrhythmia - Tachy-bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia - Tachycardia - Non-ventricular (Cardiac disorders) | 20 (21) | 1 (1)
Arrhythmia - Tachycardia - Ventricular (Cardiac disorders) | 16 (16) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 122 (122) | 10 (10)
Biliary (gallbladder) (Gastrointestinal disorders) | 2 (3) | 0 (0)
Bleeding - Cardiovascular - Major (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Bleeding - Cardiovascular - Minor (Blood and lymphatic system disorders) | 10 (10) | 0 (0)
Bleeding - Gastrointestinal lower - Minor (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Bleeding - Gastrointestinal upper - Minor (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bleeding - Genitourinary - Major (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Bleeding - Genitourinary - Minor (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Bleeding - Musculoskeletal/Dermatological - Minor (e.g. ecchymosis) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bleeding - Neurological - Major (e.g. CVA) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bleeding - Peripheral vascular - Minor (e.g. nosebleeds; hematomas) (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Bleeding - Pulmonary/Respiratory - Minor (e.g. hemothorax) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood sepsis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Blood/Lymphatic - Other (Blood and lymphatic system disorders) | 138 (159) | 14 (20)
Bone fracture/Break (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1)
Cancer - Progression of underlying disease (General disorders) | 3 (3) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 2 (2)
Cardiovascular - Other (Cardiac disorders) | 85 (95) | 13 (16)
Endocrine complications (Gastrointestinal disorders) | 6 (6) | 9 (9)
Fever - Unknown origin (General disorders) | 4 (4) | 2 (2)
Gastrointestinal - Infection (Gastrointestinal disorders) | 7 (7) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 29 (31) | 9 (9)
Genitourinary - Other (Renal and urinary disorders) | 22 (24) | 2 (2)
Hearing disorder (General disorders) | 0 (0) | 1 (1)
Heart failure - Acute (Cardiac disorders) | 65 (65) | 2 (2)
Heart Failure - Chronic (CHF) (Cardiac disorders) | 15 (15) | 1 (1)
Hepatic complication - Other (Gastrointestinal disorders) | 3 (3) | 0 (0)
Hypertension - Pulmonary (Cardiac disorders) | 2 (2) | 0 (0)
Hypertension - Systemic (Cardiac disorders) | 17 (17) | 2 (2)
Hypotension (Cardiac disorders) | 38 (40) | 14 (14)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Infection/Inflammation - Other (Musculoskeletal and connective tissue disorders) | 11 (11) | 2 (2)
Liver Failure - Chronic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Metabolic complications (Gastrointestinal disorders) | 9 (11) | 1 (1)
Muscular skeletal/Dermatologic - Other (Musculoskeletal and connective tissue disorders) | 87 (103) | 10 (12)
Nonspecific, unknown, or other body system - Other complication (General disorders) | 108 (133) | 14 (21)
NSD - Paravalvular leak +1 Minor (General disorders) | 1 (1) | 0 (0)
NSD - Paravalvular leak +2 Minor (General disorders) | 0 (0) | 2 (2)
NSD - Paravalvular leak +3 Major (General disorders) | 3 (3) | 0 (0)
Pancreatic complication (Gastrointestinal disorders) | 1 (1) | 1 (1)
Perforation - Other (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion - Minor (Cardiac disorders) | 21 (21) | 3 (3)
Pericarditis (Cardiac disorders) | 6 (6) | 1 (1)
Pleural effusion - Bilateral (Cardiac disorders) | 13 (13) | 7 (7)
Pleural effusion - Left (Cardiac disorders) | 10 (10) | 7 (7)
Pleural effusion - Right (Cardiac disorders) | 1 (1) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 31 (31) | 3 (3)
Psychiatric - Other (Psychiatric disorders) | 44 (46) | 6 (6)
Psychiatric disorder (Psychiatric disorders) | 6 (6) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 26 (26) | 3 (3)
Pulmonary embolism - Left (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism - Right (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary/Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 31 (32) | 5 (6)
Regurgitation - Aortic-central/Transvalvular +3 (Cardiac disorders) | 1 (1) | 0 (0)
Regurgitation - Mitral-central/Transvalvular +1 (Cardiac disorders) | 0 (0) | 2 (2)
Regurgitation - Mitral-central/Transvalvular +2 (Cardiac disorders) | 0 (0) | 1 (1)
Regurgitation - Mitral-central/Transvalvular +3 (Cardiac disorders) | 0 (0) | 1 (1)
Regurgitation - Mitral-central/Transvalvular +4 (Cardiac disorders) | 1 (1) | 0 (0)
Regurgitation - Mitral-indeterminate +2 (Cardiac disorders) | 2 (2) | 0 (0)
Regurgitation - Mitral-indeterminate +3 (Cardiac disorders) | 3 (3) | 0 (0)
Regurgitation - Tricuspid-indeterminate +3 (Cardiac disorders) | 1 (1) | 0 (0)
Regurgitation - Tricuspid-indeterminate +4 (Cardiac disorders) | 0 (0) | 1 (1)
Renal - Other (Renal and urinary disorders) | 18 (18) | 1 (1)
Renal dysfunction (Renal and urinary disorders) | 10 (11) | 1 (1)
Renal failure - Acute (Renal and urinary disorders) | 19 (19) | 4 (4)
Renal failure - Chronic (Renal and urinary disorders) | 2 (2) | 0 (0)
Respiratory dysfunction/Insufficiency (Respiratory, thoracic and mediastinal disorders) | 21 (21) | 1 (1)
Respiratory failure - Acute Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure - Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure - COPD (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure - Other (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 2 (3)
Respiratory failure - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Respiratory failure - Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Respiratory infection - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Respiratory infection - Upper (URI) (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 2 (2)
Speech disorder (General disorders) | 1 (1) | 1 (1)
Sternal wound/Thoracic infection (Musculoskeletal and connective tissue disorders) | 9 (9) | 0 (0)
Thrombocytopenia - Heparin Induced (HIT) (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Thrombocytopenia - Non-heparin induced (Blood and lymphatic system disorders) | 134 (134) | 18 (18)
Thromboembolic event - Stroke (Cardiac disorders) | 2 (2) | 0 (0)
Thromboembolic event - Transient Ischemic Attack (TIA) (Cardiac disorders) | 6 (6) | 0 (0)
Transient psychotic syndrome (Psychiatric disorders) | 4 (4) | 0 (0)
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 26 (26) | 6 (9)
Vascular - Access site complication (Vascular disorders) | 2 (2) | 0 (0)
Vascular - Deep Vein Thrombosis (DVT) (Vascular disorders) | 4 (4) | 1 (1)
Vascular - Other (Vascular disorders) | 19 (19) | 1 (1)
Vision disorder (General disorders) | 12 (14) | 3 (3)
Wound infection - Other (Musculoskeletal and connective tissue disorders) | 8 (8) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of overall study results which have not been released requires written approval of Sponsor, but presentation of site-specific results can occur subject to review by Sponsor. Manuscripts will be submitted to Sponsor for review 30 days prior to submission of manuscript for publication/presentation. Sponsor may ask for a 60 day delay of submission of manuscripts for publication to protect proprietary information and filing of related patent applications.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/65/NCT01757665/Prot_SAP_001.pdf